CLINICAL TRIAL: NCT07004010
Title: Evaluating the Efficacy and Safety of Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.) for the Treatment of Flank Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Espad Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB.ESP.KB.IV.02
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Flank Fat

STUDY DESIGN:
Intervention Model Description: before/after clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embella (Deoxycholic acid, produced by Espad Pharmed Co.) (Experimental)
  Interventions: Device: Deoxycholic Acid Injection

INTERVENTIONS:
Device: Deoxycholic Acid Injection — The intervention include Deoxycholic acid, SC, 0.15 ml each injection, up to 2-4 ml in each site (2 ml at visit 1 for everyone, and 2 ml at visit 2 unless the patient does not agree)

SUMMARY:
Flank region fat is a factor affecting beauty that makes people feel uncomfortable about themselves. In 2015, deoxycholic acid was approved by the American FDA for treatment of flank fat. The purpose of this study is to evaluate the efficacy and safety of deoxycholic acid injection with the brand name Embella®, manufactured by Espad Pharmed Company, for treatment of this condition.

The Primary objective of this study was the proportion of participants with grade 1 or higher ("improved, much improved, very much improved") in investigator-assessed Global Aesthetic Improvement Scale (GAIS) at Week 12 Secondary objective was assessment of other efficacy parameters as well as safety of the product

ELIGIBILITY:
Inclusion Criteria:

* Having mild to moderate flank fat assessed by the investigator and sonography and/or caliper (≥2cm thickness of the fat tissue in posterior axillary lines at the level of ASIS)
* Signing informed consent by the subject
* Ability to follow study instructions and likely to complete all required visits
* Agreement to abstain from any treatment to the flank region, including botulinum toxins, hyaluronic acid fillers, cosmetic surgery, laser/light therapy, chemical peels, etc., during the study

Exclusion Criteria:

* Planning to change lifestyle within the projected duration of the trial
* History of liposuction surgery or laser lipolysis in the past 12 months or planning to have these procedures
* Significant weight reduction in the past 6 months or planning for weight reduction within the projected duration of the trial
* BMI > 30 kg/m2
* Waist circumference > 105 cm
* Uncontrolled systemic diseases
* Severe cardiovascular diseases
* Known allergy or sensitivity to the study medication or its components
* Females who are pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study and for the duration of the study.
* Previous treatment to the flanks with hyaluronic acid fillers or semi-permanent filler in the past 12 months
* Use of any permanent filler materials or silicone in the flanks
* Subjects planning a cosmetic procedure in the treatment area during the study or with prior cosmetic procedures (i.e., surgery) in the treatment area or visible scars that may affect the evaluation
* Subjects with volume deficit due to trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disease, or HIV-related disease
* Infection or dermatoses at the injection site
* Evidence of recent alcohol or drug abuse
* Medical and/or psychiatric problems that are severe enough to interfere with the study results
* Known bleeding disorder or receiving medication that will likely increase the risk of bleeding after injection
* Having hair that would interfere with evaluation and treatment of the flank area
* Being prone to develop hypertrophic scarring
* Having a history of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), hyaluronic acid products, or Streptococcal protein
* Having porphyria
* Having an active inflammation, infection, cancerous or precancerous lesion, or unhealed wound in the flank area
* Having a condition or being in a situation that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Razi hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Flanks
Groups:
- Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.): Participants who received intervention including Deoxycholic acid, subcutaneous injection, 0.1-0.15 ml each injection, with a maximum injection volume of 2 mL per flank per session.
Period: Overall Study
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Started | 30; 60 Flanks
Completed | 30; 60 Flanks
Not Completed | 0; 0 Flanks

BASELINE CHARACTERISTICS:
Groups:
- Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.): Deoxycholic Acid Injection: The intervention included Deoxycholic acid, subcutaneous injection, 0.1-0.15 ml each injection, with a maximum injection volume of 2 mL per side per session.
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.93 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Grade 1 or Higher ("Improved, Much Improved, Very Much Improved") in Investigator-assessed Global Aesthetic Improvement Scale (GAIS) at Week 12
Description: A comparison between Week 12 and Baseline standardized photographs will be made by two independent physicians, resulting in a GAIS score from the range +3 (very much improved), +2 (much improved), +1 (improved), 0 (no change), -1 (worse), -2 (much worse), and -3 (very much worse). The average score between the investigators was taken.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
Participants | 26

2. Secondary Outcome: Safety Assessment by Evaluation of Adverse Events (AEs)
Description: Number of participants with at least one adverse event (AE). AEs were assessed at all visits.
Time Frame: Up to week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
Participants | 30

3. Secondary Outcome: The Proportion of Participants With Grade 1 or Higher ("Improved, Much Improved, Very Much Improved") in Investigator-assessed Global Aesthetic Improvement Scale (GAIS) at Week 6
Description: A comparison between Week 6 and Baseline standardized photographs will be made by two independent physicians, resulting in a GAIS score from the range +3 (very much improved), +2 (much improved), +1 (improved), 0 (no change), -1 (worse), -2 (much worse), and -3 (very much worse). The average score between the investigators was taken.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
Participants | 21

4. Secondary Outcome: Change From Baseline in Ultrasonographic Measurement of Dermal and Hypodermal Thickness on Both Flanks at Weeks 6 and 12
Time Frame: Baseline, Week 6, Week 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
mm
  Right dermis at baseline | 2.12 (0.41)
  Right dermis at week 6 | 2.27 (0.36)
  Right dermis at week 12 | 2.44 (0.42)
  Left dermis at baseline | 2.25 (0.44)
  Left dermis at week 6 | 2.44 (0.48)
  Left dermis at week 12 | 2.73 (0.49)
  Right hypodermis at baseline | 23.70 (6.35)
  Right hypodermis at week 6 | 20.87 (4.61)
  Right hypodermis at week 12 | 20.00 (3.99)
  Left hypodermis at baseline | 24.68 (6.43)
  Left hypodermis at week 6 | 22.25 (4.96)
  Left hypodermis at week 12 | 20.69 (4.46)
Statistical Analysis 1: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); This statistical analysis pertains to the right dermis and evaluates the trend across baseline, Week 6, and Week 12; Test type: Other; p < 0.001, Friedman
Statistical Analysis 2: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); This statistical analysis pertains to the left dermis and evaluates the trend across baseline, Week 6, and Week 12; Test type: Other; p < 0.001, Friedman
Statistical Analysis 3: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); This statistical analysis pertains to the right hypodermis and evaluates the trend across baseline, Week 6, and Week 12; Test type: Other; p < 0.001, Repeated measure

5. Secondary Outcome: Changes From Baseline in the Bodyweight (Kg) at Weeks 6 and 12
Time Frame: Baseline, Week 6, Week 12
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
Kg
  Baseline | 68.57 (9.32)
  Week 6 | 68.90 (9.49)
  Week 12 | 69.13 (9.24)
Statistical Analysis 1: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Test type: Other; p = 0.264, Repeated measure

6. Secondary Outcome: Changes From Baseline in Right and Left Thigh Circumference at Weeks 6 and 12 Using a Flexible Tape Measure
Time Frame: Baseline, Week 6, Week 12
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
cm
  Right thigh at baseline | 59.98 (3.65)
  Right thigh at week 6 | 59.82 (3.87)
  Right thigh at week 12 | 60.23 (3.37)
  Left thigh at baseline | 59.50 (3.74)
  Left thigh at week 6 | 59.03 (3.82)
  Left thigh at week 12 | 59.35 (3.75)
Statistical Analysis 1: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Right thigh; Test type: Other; p = 0.278, Repeated measure
Statistical Analysis 2: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Left thigh; Test type: Other; p = 0.061, Repeated measure

7. Secondary Outcome: Changes From Baseline in Caliper Measurement (mm) of Flank Fat on Each Side at Weeks 6 and 12
Time Frame: Baseline, Week 6, Week 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
mm
  Right caliper at baseline | 4.89 (0.58)
  Right caliper at week 6 | 4.52 (0.62)
  Right caliper at week 12 | 4.16 (0.59)
  Left caliper at baseline | 4.76 (0.59)
  Left caliper at week 6 | 4.43 (0.60)
  Left caliper at week 12 | 4.03 (0.56)
Statistical Analysis 1: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Right caliper; Test type: Other; p < 0.001, Repeated measure
Statistical Analysis 2: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Left caliper; Test type: Other; p < 0.001, Repeated measure

8. Secondary Outcome: Changes From Baseline in Waist Circumference at Weeks 6 and 12 Using a Flexible Tape Measure
Time Frame: Baseline, Week 6, Week 12
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
cm
  Baseline | 91.83 (6.66)
  week 6 | 90.72 (6.31)
  week 12 | 88.98 (6.20)
Statistical Analysis 1: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Test type: Other; p < 0.001, Repeated measure

9. Secondary Outcome: Subject's Satisfaction at Weeks 6 and 12 Using a 10-point Likert Scale
Description: A 10-point Likert scale is used to measure subject's satisfaction, comprising a question followed by a scale with ten choices, going from "1" (Completely dissatisfied) to "10" (Completely satisfied).
Time Frame: Week 6, Week 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
Number analyzed (Participants) | 30
score on a scale
  week 6 | 7.0 [6.0 to 8.0]
  week 12 | 7.5 [5.0 to 9.0]
Statistical Analysis 1: Comparison: Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.); Test type: Other; p = 0.894, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline, Week 6, Week 12
Arm/Group | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 30/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Embella (Deoxycholic Acid, Produced by Espad Pharmed Co.) (N=30)
Injection site bruising (General disorders) | 26
Injection site pain (General disorders) | 21
Injection site swelling (General disorders) | 10
Injection site pruritus (General disorders) | 8
Injection site necrosis (General disorders) | 1
injection site urticaria (General disorders) | 1
injection site skin tightness (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT07004010/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT07004010/SAP_001.pdf